CLINICAL TRIAL: NCT04018040
Title: Efficacy of a Lacto-ovo Vegetarian Diet in Mild to Moderate IBD
Brief Title: Vegetarian Diet in IBD
Acronym: LOVIBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edith Cowan University (Other)
Collaborators: St John of God Healthcare, Perth (Unknown); Fiona Stanley Fremantle Hospitals Group (Unknown); Royal Perth Hospital (Other)
Responsible Party: Principal Investigator, Charlene Grosse, Advanced Accredited Practising Dietitian, PhD Candidate, Edith Cowan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EdithCowanU
Record Dates: First submitted 2019-05-26; First posted 2019-07-12 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Ulcerative Colitis; Crohn Disease; Inflammatory Bowel Diseases
Keywords: Diet; Plant based diet; Lacto ovo vegetarian diet
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases | interventions — Diet, Vegetarian

STUDY DESIGN:
Intervention Model Description: Phase 1: Open labelled, single centre trial in mild to moderate UC ( n=14) Phase 2:Open labelled, single centre trial in mild to moderate CD (n-12)
Masking Description: Due to the nature of this type of dietary intervention it is not possible to blind the participant nor treating gastroenterolgist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Patients will follow a lacto-ovo vegetarian diet for an 8 week period. patients will be provided with a lacto-ovo vegetarian food box delivery service with fresh ingredients and recipes to cover four dinners per week.
  Interventions: Other: Lacto-ovo vegetarian diet

INTERVENTIONS:
Other: Lacto-ovo vegetarian diet — Lacto-ovo vegetarian diet inclusive of dairy and eggs

SUMMARY:
To determine whether a lacto-ovo vegetarian diet is effective in improving gastrointestinal symptoms, quality-of-life, intestinal inflammation and gut microbiota composition in mild-to-moderate IBD compared to a standard omnivorous diet.

DETAILED DESCRIPTION:
This study will review whether a lacto-ovo vegetarian diet is an optimal dietary therapy to achieve a clinical response in mild to moderate UC and CD as an adjunctive treatment to current medical therapies. The proposed studyT will be used to evaluate the efficacy of a lacto-ovo vegetarian diet together with its effect on the microbiota to create an enhanced understanding of the role diet plays in the management midl to moderate IBD. Using a socially acceptable diet it is anticipated that food-related quality-of-life measures will improve for participants. Dietary modification could be a more economical, safer and more effective means of reducing symptoms and flare-ups compared to pharmacological therapy.

ELIGIBILITY:
Inclusion Criteria I. Is able to provide informed consent. II. Is over the age of 18 years. III. Has a diagnosis of ulcerative colitis or Crohn's disease for over a 3-month duration that was confirmed by a specialist gastroenterologist IV. Pro-6 score of 2 to 4, partial mayo 3-6 (mild to moderate UC) or Harvey Bradshaw Index (HBI) 5 to 15 (Crohn's disease)

V. Medications:

1. Oral 5-Aminosalicylates: If taking an oral 5-Aminosalicylates the patient has used them continuously for 4 weeks and has been on a stable dose for 2 weeks prior to the screening visit.
2. Oral Corticosteroids: If taking oral corticosteroids the patient has used them continuously for 4 weeks and has been on a stable dose for 2 weeks prior to the screening visit at a dose of ≤30mg.
3. Oral Azathioprine/6MP, Methotrexate or tacrolimus: If taking one of these medications the patient has used them for a minimum of 12 weeks and has been on a stable dose for 4 weeks prior to screening.
4. Biologic therapy with infliximab, adalimumab or vedolizumab: If taking one of these medications the patient has used them for a minimum of 12 weeks
5. Rectal Preparations; 5-Aminosalicylates, corticosteroids or tacrolimus: If taking one of these medications the patient has used them continuously for 4 weeks and has been on a stable dose for 2 weeks prior to the screening visit.

VI. Willing to participate in the study and comply with the proceedings by signing a written informed consent.

VII. Free of any clinically significant disease, other than ulcerative colitis/Crohn's disease, that would interfere with the study's evaluations.

VIII. Subjects can read and understand English and is able to adhere to the study methodology and visit schedules.

Exclusion Criteria

I. Has been on antibiotics within the last four weeks. II. Has a known food allergy to nuts, soy, eggs or dairy. III. Is pregnant or breast feeding. IV. Following a vegetarian, vegan or low FODMAP diet. V. Has known dementia and the inability to understand the trial requirements. VI. Ulcerative colitis: Patients with less than 15cm of disease (proctitis) VII. Crohn's disease: Patients with severe Disease (HBI > 15) or remission (HBI<5) VIII. Patients with active extraintestinal disease, current B2 (Fixed non inflammatory stricture1 or small bowel obstruction) or B3 disease (Boneh et al, 2017)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with a clinical response at week 8 | Week 8
  A clinical response is defined as a decrease from baseline in the total Mayo score of at least three points, with an accompanying decrease in the subscore for rectal bleeding or at least 1 point or an absolute subscore for rectal bleeding of 0 or 1

SECONDARY OUTCOMES:
Number of participants achieving clinical remission at week 8 | Week 8
  A clinical remission is defined by a total Mayo score of 2 points or lower, with no individual subscore exceeding 1 point or a reduction in HBI of three points
Number of participants with changes to IBDQ score at week 8 | Week 8
  Change in total score from baselines. IBDQ - normal quality of life score is 170 points (range 32 to 224) and a quality of life response is a change of 16 points.
Participants Food related quality of life in IBD (Fr-QoL 29) score at week 8 | Week 8
  Change in total score from baseline. Lowest score of 29 reflects poor quality of life, maximum score of 145 reflects highest quality of life score.
Participants SF-36 quality of life score at week 8 | Week 8
  SF-36- change in total score from baseline. A score of 0 reflects maximum disability, the maximum score of 100 reflects no disability.
Number of participants achieving a change in gut microbiome diversity at week 8 | Week 8
  The gut microbiome will be examined using ITS2, 16S rRNA gene and metagenomics.
Number of participants with a change in beneficial gut metabolome profile at week 8 | Week 8
  Untargeted metabolomics will be performed on stool samples using high-resolution Gas Chromatography Mass Spectrometry (GC-Orbitrap-MS). Metabolite identification will be established prior to statistical analysis, by matching against an in-house MS/MS spectral library of 900 metabolites and searching online spectral libraries (mzCloud, Metlin, HMDB and Massbank).

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Liverpool Hospital, Sydney, New South Wales
  - St John of God Subiaco Hospital, Perth, Western Australia
  - Fiona Stanley Fremantle Hospitals Group, Perth, Western Australia
  - Royal Perth Hospital, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No
All data will be de-identified

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-11-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT04018040/Prot_SAP_ICF_001.pdf